CLINICAL TRIAL: NCT02761941
Title: Excessive Warfarin Anticoagulation - Causes and Consequences
Acronym: EWA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor of Cardiology, University of Turku
Other Study IDs: T80/2016
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the clinical significance of high INR (International Normalized Ratio) values (>9) in VKA (vitamin K antagonist) treated patients with atrial fibrillation. The clinical characteristics of these patients will be studied as well as the clinical presentation. Factors influencing on high INR values will be recorded and the aim is to seek out patients who have elevated risk of bleeding complications.

DETAILED DESCRIPTION:
This is a retrospective study setting. Source data will be collected by reviewing medical records and through computer searches. The basic study population will be identified from laboratory INR test results taken between 2003-2015.

Identifying patients with INR values over 9 will be selected for further analysis, concerning the clinical presentation, patient characteristics, 90 day survival and adverse event rates. The focus is in identifying patient characteristics and factors influencing the risk of high INR value. Also we will analyse the effects of medically reversing the high INR values on stroke and other adverse event rates. The results will be collected manually using an electronic case report form, and analysed statistically using SPSS/SAS statistics tool.

ELIGIBILITY:
Inclusion Criteria:

* VKA treatment, age > 18, INR >9,

Exclusion Criteria:

* age < 18

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with VKA for atrial fibrillation in the Southwest Finland hospital district area with INR value over 9.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Airaksinen, Professor, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided